CLINICAL TRIAL: NCT06014606
Title: How Does the Brain Learn About Positive and Negative Things?
Brief Title: Learning and Decision-making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DANE1
Record Dates: First submitted 2022-09-05; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Motivation
MeSH Terms: interventions — Haloperidol; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind (randomised) between-subjects design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HV/Placebo (Placebo Comparator): Oral placebo (tablet)
  Interventions: Drug: placebo
- HV/Haloperidol (Active Comparator): 2mg (oral)
  Interventions: Drug: haloperidol 2mg
- HV/Propranolol (Active Comparator): 40mg (oral)
  Interventions: Drug: propranolol 40mg

INTERVENTIONS:
Drug: placebo — oral formulation
  Arms: HV/Placebo
Drug: haloperidol 2mg — oral formulation
  Arms: HV/Haloperidol
Drug: propranolol 40mg — oral formulation
  Arms: HV/Propranolol

SUMMARY:
A fundamental aspect of daily life decision-making involves the evaluation of costs and benefits. Neural systems underlying cost-benefit evaluation have been extensively examined, but the specific role of different neurotransmitters remains unclear. Numerous studies suggest that both dopamine (DA) and norepinephrine (NE) are closely related to reinforcement learning, guided exploration/exploitation, and behavioural energisation, although no studies to date have investigated the distinct role of DA and NE on cost-benefit decision-making and learning in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Age between 18 and 35
* Body-Mass Index (BMI) between 17.5-30
* Availability for participation through the duration of the study

Exclusion Criteria:

* Diagnosis of a psychiatric or neurological disorder, including substance abuse or dependence (yes/no self-report - lifetime)
* Use of any psychopharmacological treatment 3 weeks before the test day (yes/no self-report)
* Use of any blood pressure medication (yes/no self-report - lifetime)
* Pregnancy (confirmed via urine pregnancy test) or nursing (yes/no self-report) or have plans to get pregnant in the near future (yes/no self-report) (females only)
* Diagnosis of a cardiac disease (medical questionnaire), obstructive respiratory disease (medical questionnaire), abnormal blood pressure (diastolic< 60mmHg; systolic< 90mmHg) (medical screening)
* Chronic renal failure (medical questionnaire)
* Hypothyroidism (medical questionnaire)
* Diabetes (medical questionnaire)
* Hypersensitivity to phenothiazines (medical questionnaire)
* Diagnosis of a cardiac disease (medical questionnaire)
* Alcohol consumption in the 24 hours before the test session starts (yes/no self-report)
* Food intake less than 3 hours before the test day (yes/no self-report)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Cost-benefit reinforcement learning performance | ~ 2.5 hours post-drug administration
  2-choice reinforcement learning task (based on Voulgaropoulou et al., 2021 PNEC)

SECONDARY OUTCOMES:
Effort-based decision-making | ~ 2 hours post-drug administration
  motivation to acquire rewards (e.g., Reddy et al. 2015)

OTHER OUTCOMES:
Physiology I | pre, +30 min., +60 min., +90 min., +120 min., +190 min. post-drug administration
  Heart rate
Physiology II | pre, +30 min., +60 min., +90 min., +120 min., +190 min. post-drug administration
  blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Voulgaropoulou SD, Fauzani F, Pfirrmann J, Vingerhoets C, van Amelsvoort T, Hernaus D. Asymmetric effects of acute stress on cost and benefit learning. Psychoneuroendocrinology. 2022 Apr;138:105646. doi: 10.1016/j.psyneuen.2021.105646. Epub 2021 Dec 24. PMID 35065334